CLINICAL TRIAL: NCT01130051
Title: A Pilot Bioavailability Study of Colcrys® Tablet 0.6 mg Versus Colcrys® Tablets 0.6 mg Crushed and Sprinkled on Applesauce Under Fasting Conditions
Brief Title: Bioavailability Study of Colcrys® Crushed and Sprinkled on Applesauce
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Medical Director, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-10-1002
Record Dates: First submitted 2010-05-21; First posted 2010-05-25 (Estimated); Results first posted 2011-05-11 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: bioavailability
MeSH Terms: interventions — Colchicine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colcrys® 0.6 mg intact tablet (Experimental): One Colcrys® 0.6 mg intact tablet taken by mouth
  Interventions: Drug: Colchicine 0.6 mg tablet
- Colcrys® 0.6 mg tablet on applesauce (Experimental): One Colcrys® 0.6 mg tablet crushed and sprinkled on applesauce
  Interventions: Drug: Colchicine 0.6 mg tablet

INTERVENTIONS:
Drug: Colchicine 0.6 mg tablet — One Colcrys® 0.6 mg intact tablet taken by mouth
  Other Names: Colcrys®
  Arms: Colcrys® 0.6 mg intact tablet
Drug: Colchicine 0.6 mg tablet — One Colcrys® 0.6 mg tablet crushed and sprinkled on applesauce
  Other Names: Colcrys®
  Arms: Colcrys® 0.6 mg tablet on applesauce

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability of a single 0.6 mg tablet of Colcrys® (colchicine, USP) when crushed and sprinkled on applesauce (1 tablespoon) relative to the same dose given as an intact tablet to healthy subjects following an overnight fast. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability of a single 0.6 mg tablet of Colcrys® (colchicine, USP) when crushed and sprinkled on applesauce (1 tablespoon) relative to the same dose given as an intact tablet to healthy subjects following an overnight fast. Sixteen healthy, non-smoking, non-obese, male and female volunteers between 18-55 years of age will be randomly assigned in a crossover fashion to receive each of two dosing regimens in sequence with a 14 day washout period between dosing periods. In each of the dosing periods, after an overnight fast, subjects will receive one intact Colcrys® 0.6 mg tablet (followed by 240 mL of water) or one Colcrys® 0.6 mg tablet crushed and sprinkled on 1 tablespoon of applesauce (followed by 240 ml of water) according to the randomization schedule. Blood samples will be drawn from all participants before dosing and for 48 hours post-dose at times sufficient to adequately define the pharmacokinetics of colchicine. Vital signs (blood pressure, heart rate, respiratory rate and temperature) will be measured prior to dosing, 1 hour ± 30 minutes post-dose and upon discharge from the clinical facility. Subjects will be monitored throughout their participation in the study for adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults age 18-55, non-smoking, non- pregnant (post-menopausal, surgically sterile or using effective contraceptive measures) with a body mass index of 18-30 kg/m²

Exclusion Criteria:

* Recent participation (within 30 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* History of treatment for drug or alcohol addiction within the previous 12 months or use of tobacco products within 90 days of the start of the study
* Significant history or current evidence of chronic infectious disease, system disorders, organ dysfunction, especially cardiovascular disorders (angina, heart failure, irregular heartbeats, heart attack, hypertension, hypotension) stroke, renal or hepatic disorders, diabetes or bleeding disorders, gastrointestinal disease or history of malabsorption within the last year
* History of psychiatric disorders occurring within the last two years that required hospitalization or medication
* Presence of a medical condition requiring regular treatment with prescription drugs
* Use of any drugs or substances known to inhibit or induce drug-metabolizing enzymes within 30 days prior to dosing with the study drug
* Drug allergies or sensitivity to colchicine
* Positive test results for drugs of abuse at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, M.D., Study Chair — Mutual Pharmaceutical Company, Inc.
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Colcrys® Intact Tab Then Colcrys® Sprinkled on Applesauce: On the morning of Day 1, subjects received the reference formulation, one intact tablet of Colcrys® 0.6 mg after an overnight fast of at least 10 hours. Following a 14 day washout period, on the morning of Day 15, subjects received the test formulation, one Colcrys® 0.6 mg tablet crushed and sprinkled on applesauce, after an overnight fast of at least 10 hours
- Colcrys® Sprinkled on Applesauce Then Colcrys® Intact Tab: On the morning of Day 1 subjects received one tablet of the test formulation, Colcrys® 0.6 mg, crushed and sprinkled on applesauce, after an overnight fast of at least 10 hours. Following a 14 day washout period, on the morning of Day 15, subjects received one dose of the reference formulation, one intact Colcrys® 0.6 mg tablet, after an overnight fast of at least 10 hours
Period: Period 1
Arm/Group | Colcrys® Intact Tab Then Colcrys® Sprinkled on Applesauce | Colcrys® Sprinkled on Applesauce Then Colcrys® Intact Tab
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout Period of 14 Days
Arm/Group | Colcrys® Intact Tab Then Colcrys® Sprinkled on Applesauce | Colcrys® Sprinkled on Applesauce Then Colcrys® Intact Tab
Started | 8 | 8
Completed | 7 | 6
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 1
Period: Period 2
Arm/Group | Colcrys® Intact Tab Then Colcrys® Sprinkled on Applesauce | Colcrys® Sprinkled on Applesauce Then Colcrys® Intact Tab
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Colcrys® Intact Tab and Colcrys® in Applesauce: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 15, each subject received one tablet of intact Colcrys® 0.6 mg or one tablet of Colcrys® 0.6 mg crushed and sprinkled on applesauce, following an overnight fast of at least 10 hours.
Arm/Group | Colcrys® Intact Tab and Colcrys® in Applesauce
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.812 (13.332)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that Colcrys® reaches in the plasma
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 16, 18, 20, 24, 36, and 48 hours after drug administration
Population: Plasma concentration data for 13 of 16 participants were used in the statistical analysis. One subject dropped from the study before Period 2 dosing for personal reasons. Two subjects were discontinued from the study before Period 2 for protocol violations.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Colcrys® 0.6 mg Administered as an Intact Tablet: Each subject received one intact tablet of Colcrys® 0.6 mg after an overnight fast of at least 10 hours
- Colcrys® 0.6 mg Tablet Crushed and Sprinkled on Applesauce: Each subject received one tablet of Colcrys® 0.6 mg crushed and sprinkled on applesauce after an overnight fast of at least 10 hours
Arm/Group | Colcrys® 0.6 mg Administered as an Intact Tablet | Colcrys® 0.6 mg Tablet Crushed and Sprinkled on Applesauce
Number analyzed (Participants) | 13 | 13
ng/mL | 3.087 (0.953) | 2.616 (0.785)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable Colcrys® concentration (t), as calculated by the linear trapezoidal rule
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Colcrys® 0.6 mg Administered as an Intact Tablet | Colcrys® 0.6 mg Tablet Crushed and Sprinkled on Applesauce
Number analyzed (Participants) | 13 | 13
ng-hr/mL | 23.042 (6.100) | 19.216 (4.512)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC (0-∞) was calculated as the sum of AUC (0-t) plus the ratio of the last measurable Colcrys® plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Colcrys® 0.6 mg Administered as an Intact Tablet | Colcrys® 0.6 mg Tablet Crushed and Sprinkled on Applesauce
Number analyzed (Participants) | 13 | 13
ng-hr/mL | 28.550 (8.597) | 23.883 (6.102)

ADVERSE EVENTS:
Description: One subject withdrew voluntarily from the study and one was discontinued for protocol violations after receiving the test formulation. One subject was discontinued for protocol violations after receiving the reference formulation.
Groups:
- Colcrys® 0.6 mg Tablet Administered Intact; Colcrys® 0.6 mg Tablet Crushed and Sprinkled on Applesauce: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 15, each subject received one intact tablet of Colcrys® 0.6 mg or one tablet of Colcrys® 0.6 mg crushed and sprinkled on applesauce, following an overnight fast of at least 10 hours.
Arm/Group | Colcrys® 0.6 mg Tablet Administered Intact | Colcrys® 0.6 mg Tablet Crushed and Sprinkled on Applesauce
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colcrys® 0.6 mg Tablet Administered Intact (N=14) | Colcrys® 0.6 mg Tablet Crushed and Sprinkled on Applesauce (N=15)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days